CLINICAL TRIAL: NCT01357031
Title: Double Blind Randomized Study Controlled by Placebo and Amitriptylin to Evaluate the Efficacy of Melatonin in the Preventive Treatment of Migraine
Brief Title: Study With Amitriptylin to Evaluate the Efficacy of Melatonin in Treatment of Migraine
Acronym: EDUMAP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Mario Fernando Pietro Peres, PhD, Hospital Israelita Albert Einstein
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EDUMAP
Record Dates: First submitted 2010-05-14; First posted 2011-05-20 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Migraine
Keywords: Amitriptyline; Placebo; Melatonin; Migraine; Headache; Drug therapy; Preventive treatment of migraine
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — Amitriptyline; Melatonin

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Melatonin (Experimental): Melatonin 3 mg at bedtime
  Interventions: Drug: Melatonin
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Amitriptyline (Active Comparator): Amitriptyline 25 mg
  Interventions: Drug: Amitriptyline

INTERVENTIONS:
Drug: Amitriptyline — It will be administered Amitriptyline (25mg) once a day at bed time. Patients may keep their abortive treatment that they usually used. The drug will be encapsulated in a bottle of 30 capsules will be given to patients at every visit.
  Arms: Amitriptyline
Drug: Melatonin — It will be administered Melatonin (3mg) at bed time, half an hour before the usual time of sleep of the patient.
  Arms: Melatonin
Drug: Placebo — It will be administered placebo capsules, identical to Melatonin (3mg) and Amitriptyline (25 mg) patients will take the study medication at bed time
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effectiveness of melatonin 3 mg compared to placebo and amitriptyline 25 mg in the preventive treatment of migraine.

DETAILED DESCRIPTION:
The investigators propose a study of patients with migraine (episodic) with or without aura, according to the criteria of the International Headache Society (IHS) 2004. This will be a randomized clinical trial, prospective, double-blind, placebo-controlled, comparing the efficacy of melatonin 3 mg and amitriptyline 25 mg for migraine prevention. The length of the inclusion of the study will be 24 months. This study's general objective is: to evaluate the effectiveness of melatonin in the preventive treatment of migraine and compare it to placebo and amitriptyline.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman 18 to 65 years of age.
* Meets diagnostic criteria criteria of International Headache Society (IHS) 2004 (2) for migraine with and / or without aura.
* Frequency from 2 to 8 migraine attacks per month
* Top of crisis over a year and age of onset less than 50 years of age.
* Patients want to participate in the study, and able to give informed consent.
* If women, the patient must be willing to use an acceptable method of birth control (eg, a hormonal contraceptive, intrauterine device, diaphragm with spermicide or condom with spermicide, or refer abstinence).
* Patient able and willing to remain on their medications throughout the study.
* Accept the guidelines of the study by filling out the diary and clinical scales.

Exclusion Criteria:

* Any medical condition that places the patient at risk with its exposure to melatonin or amitryptiline
* Use of alcohol and drugs.
* Be receiving prophylactic medication in the last three months.
* History of hemiplegic migraine, basilar, Ophthalmoplegic or stroke.
* Headache secondary to head trauma or a whiplash neck injury (whiplash).
* Pregnant or breastfeeding. Women planning to become pregnant or of childbearing age without acceptable method of contraception.
* Women who began taking oral contraceptives or who switched their oral contraceptive regimen in the 6 months prior to the start of the study.
* Allergy or known hypersensitivity to study medication or its components.
* Participation in another clinical study one month before inclusion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2010-05; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change in number of headache days from baseline to month 3 after treatment. | Baseline (4 weeks) and treatment period (12 weeks)
  This is a randomized, double-blind, placebo-controlled, parallel-group, multicenter study to evaluate the efficacy of melatonin 3 mg, amitriptyline 25 mg versus placebo in the prevention of migraine headaches. The study consists of 2 phases: Baseline Phase (4 weeks) and Double-Blind Phase (patients are randomized to receive melatonin, amitriptyline or placebo for a total of 12 weeks).

SECONDARY OUTCOMES:
Proportion of patients responding to treatment. Change from Baseline Phase to Double-Blind Phase in number of monthly migraine attacks, migraine intensity, migraine duration, analgesic use, weight (in kg), and tolerability reports. | Baseline (4 weeks) and treatment period (12 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Mario F Peres, PhD, Principal Investigator — Hospital Israelita Albert Einstein
Locations (1):
- Instituto Israelita de Ensino e Pesquisa Albert Einstein, São Paulo, São Paulo, Brazil